CLINICAL TRIAL: NCT06417528
Title: Chronic Postsurgical Pain: Multivariate Prediction Model
Acronym: CPoP
Status: Recruiting | Type: Observational
Sponsor: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, Luigi Cardia, Principal Investigator, Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva
Other Study IDs: CPoP
Record Dates: First submitted 2024-03-19; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Post Surgical Pain; Post Operative Pain; Postoperative Pain, Chronic
Keywords: Pain; Chronic Pain; Postoperative Pain; Post Operative Pain; Post Surgical Pain; Multivariate Prediction Model; Prediction Model
MeSH Terms: conditions — Pain, Postoperative; Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery Patients: Data collection will record parameters of patients undergoing surgery at four different times: preoperative assessment (60 to 1 day before the scheduled procedure); evaluation of the perioperative period; and postoperative period (from the third month following surgery).
  Interventions: Procedure: Chronic Post Surgery Pain (CPSP)

INTERVENTIONS:
Procedure: Chronic Post Surgery Pain (CPSP) — The outcome variable is the presence of CPSP assessed 3 months after surgery and defined as an average pain intensity of at least 3 on the NRS scale (11-point one-dimensional pain scale) in the last three days, and pain localized to the surgical field (or in the lesion area) projected into the innervation territory of a nerve located in this area or referred to a dermatome.
  Separate prediction models will be developed using data derived from surveys conducted at the relevant time points for the development of the risk index.

SUMMARY:
The goal of this observational study is to identify the risk factors of Chronic Postoperative pain (or Chronic Post Surgery Pain - CPSP) three months after surgery and, subsequently. the development of a risk index to identify high-risk patients considering the multifactorial etiology of CPOP in adult patients undergoing any type of elective surgery.

DETAILED DESCRIPTION:
The study aims to identify the risk factors of CPSP three months after surgery and subsequently develop a risk index to identify high-risk patients considering the multifactorial etiology of CPSP.

A comprehensive entry pool was derived from a systematic literature search. Data collection will record parameters at four different time points: preoperative assessment (60 to 1 day before the scheduled procedure); evaluation of the perioperative period; postoperative period (from the third month after the operation).

The outcome variable is the presence of CPSP assessed 3 months postoperatively and defined as a mean pain intensity of at least 3 on the NRS (one-dimensional pain scale from 0 to 10) over the past three days and pain localized to the field surgical (or to the area of the lesion) projected into the innervation territory of a nerve located in this area, or referred to a dermatome.

Four separate forecasting models will be developed using data derived from surveys carried out at relevant time points for the development of the risk index.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Patients undergoing any type of elective surgery

Exclusion Criteria:

* Patients with sensory impairments
* Patients unable to communicate
* Patients with cognitive impairments
* Patients with insufficent knowledge of the language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing any type of elective surgery
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Chronic Post Surgery Pain (CPSP) | 3 months
  Presence of CPSP assessed 3 months after surgery and defined as an average pain intensity of at least 3 points on the NRS scale (one-dimensional pain scale - from 0 to 10 points) in the last three days and pain localized to the surgical field (or in the lesion area) projected into the innervation territory of a nerve located in this area, or referred to a dermatome.

SECONDARY OUTCOMES:
Pre operative factors | 60 to 1 day before the scheduled procedure
  * Age
    * 18-35
    * 36-55
    * ≥55
  * Sex
    * Female
    * Male
  * BMI
    * ≤18.5 - 24.9
    * 25 - 29.9
    * ≥30
  * Alcohol or substances of abuse (Y/N) (specify the substance)
  * Previous experience of pain NRS ≥5 for 7 days (Y/N)
  * Presence of chronic pathologies (Y/N) (if yes, provide the list of medications)
  * Pharmacological treatments including supplements or nutraceuticals (continuous in the last 3 months) (Y/N) (if yes, provide the list of drugs)
  * Chronic pain (NRS ≥3 for ≥3 months) (Y/N)
  * Neuropathic pain (Y/N) (assessment using Douleur Neuropathique en 4 questions DN-4 questionnaire)
  * Pain catastrophizing (Y/N) (assessment via Pain Catastrophizing Scale PCS questionnaire)
  * Anxiety (Y/N) (assessment using General Anxiety Disorder-7 GAD-7 questionnaire)
  * Depression (Y/N) (assessment using Beck Depression Inventory BDI-II questionnaire)
  * Presence of pain in the last three days (NRS ≥3 mean pain intensity in the 24 hours) (Y/N)
Perioperative factors - before surgery | The day of the scheduled surgery - before the surgery
  * Site of surgery
    * Head
    * Vertebral column
    * Arms/legs
    * Chest
    * Abdomen
    * Genitourinary system
  * Surgical technique
    * Open surgery
    * Minimally invasive surgery
    * Robotic surgery
  * ERAS (enhanced recovery after surgery) protocol (Y/N)
  * Anesthesiologic technique
    * General Anesthesia
    * Spinal Anesthesia
    * Epidural Anesthesia
    * Peripheral nerve block
  * Preventive/protective analgesia (Y/N)
  * Premedication (Y/N)
  * OFA opioid-free anesthesia protocol (Y/N)
  * Postoperative analgesic prescription (Y/N)
Perioperative factors - after surgery | Immediately after the surgery to 48 hours after the surgery
  * Pain NRS score ≥3 at the end of the surgery (Y/N)
  * Presence of pain (NRS ≥5 - average value in the 24 hours) in the region of the operation at rest or during movement after surgery (Y/N)
  * Analgesic prescription after surgery
    * ≤12 hours of coverage
    * 13-24 hours of coverage
    * ≥ 24 hours of coverage
  * Postoperative surgical complications (Y/N)
  * Postoperative infectious complications (Y/N)
  * Mobilization after surgery ≤6 hours? (Y/N)
Post operative factors | 3 months after surgery
  * Pain assessment: average pain intensity assessed using a standard NRS scale (the cutoff score will be set at ≥3 mean pain intensity over the last three days ) (Y/N).
  * Diagnosis of CPSP (the pain is localized in the surgical field or in the area of the lesion, projected into the innervation territory of a nerve located in this area, or referred to a dermatome) (Y/N)
  * Surgical complications (Y/N)
  * Infectious complications related to surgery (Y/N)
  * Malignancy (Y/N)
  * Neuropathic pain (Y/N) (assessed using Douleur Neuropathique in 4 questions DN-4 questionnaire)

OTHER OUTCOMES:
Development of the risk index | 6 months after the primary completion of the study
  * Primary version of the risk index, made up of items derived from a systematic bibliographic search (compilation of the item pool).
  * Authors will analyze the associations between each of these indices and the probability of CPSP 3 months after surgery (dichotomous variable), evaluated using logistic regression models.
  * Items that were found to be significant in the bivariate analyses will then be analyzed multivariately (logistic regression models).
  * Authors will safeguard the results of the multivariate analyses by calculating the area under the ROC curve of the model, and then, the cut-off score for a high risk of developing CPSP will be identified with an optimal compromise between sensitivity and specificity.
  * The items that will generate significant predictive factors in the logistic regression analyses will be collected into an index. For each value of this index, the Authors will calculate the proportion of patients who reported CPSP at 3 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU G. Martino, Messina, Italy

REFERENCES:
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Goldberg DS, McGee SJ. Pain as a global public health priority. BMC Public Health. 2011 Oct 6;11:770. doi: 10.1186/1471-2458-11-770. PMID 21978149
- [Background] Phillips CJ. Economic burden of chronic pain. Expert Rev Pharmacoecon Outcomes Res. 2006 Oct;6(5):591-601. doi: 10.1586/14737167.6.5.591. PMID 20528505
- [Background] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Background] Turk DC, Fillingim RB, Ohrbach R, Patel KV. Assessment of Psychosocial and Functional Impact of Chronic Pain. J Pain. 2016 Sep;17(9 Suppl):T21-49. doi: 10.1016/j.jpain.2016.02.006. PMID 27586830
- [Background] Gerbershagen HJ, Dagtekin O, Rothe T, Heidenreich A, Gerbershagen K, Sabatowski R, Petzke F, Ozgur E. Risk factors for acute and chronic postoperative pain in patients with benign and malignant renal disease after nephrectomy. Eur J Pain. 2009 Sep;13(8):853-60. doi: 10.1016/j.ejpain.2008.10.001. Epub 2008 Nov 14. PMID 19010073
- [Background] Mathes T, Pape-Kohler C, Moerders L, Lux E, Neugebauer EAM. External Validation and Update of the RICP-A Multivariate Model to Predict Chronic Postoperative Pain. Pain Med. 2018 Aug 1;19(8):1674-1682. doi: 10.1093/pm/pnx242. PMID 29121211
- [Background] Althaus A, Hinrichs-Rocker A, Chapman R, Arranz Becker O, Lefering R, Simanski C, Weber F, Moser KH, Joppich R, Trojan S, Gutzeit N, Neugebauer E. Development of a risk index for the prediction of chronic post-surgical pain. Eur J Pain. 2012 Jul;16(6):901-10. doi: 10.1002/j.1532-2149.2011.00090.x. Epub 2011 Dec 23. PMID 22337572
- [Background] Sangesland A, Storen C, Vaegter HB. Are preoperative experimental pain assessments correlated with clinical pain outcomes after surgery? A systematic review. Scand J Pain. 2017 Apr;15:44-52. doi: 10.1016/j.sjpain.2016.12.002. Epub 2016 Dec 19. PMID 28850344
- [Background] Siao P, Cros DP. Quantitative sensory testing. Phys Med Rehabil Clin N Am. 2003 May;14(2):261-86. doi: 10.1016/s1047-9651(02)00122-5. PMID 12795516
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Werner MU, Mjobo HN, Nielsen PR, Rudin A. Prediction of postoperative pain: a systematic review of predictive experimental pain studies. Anesthesiology. 2010 Jun;112(6):1494-502. doi: 10.1097/ALN.0b013e3181dcd5a0. PMID 20460988
- [Background] Abrishami A, Chan J, Chung F, Wong J. Preoperative pain sensitivity and its correlation with postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2011 Feb;114(2):445-57. doi: 10.1097/ALN.0b013e3181f85ed2. PMID 21245740
- [Background] Kuner R, Flor H. Structural plasticity and reorganisation in chronic pain. Nat Rev Neurosci. 2016 Dec 15;18(1):20-30. doi: 10.1038/nrn.2016.162. PMID 27974843
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Campos ACP, Antunes GF, Matsumoto M, Pagano RL, Martinez RCR. Neuroinflammation, Pain and Depression: An Overview of the Main Findings. Front Psychol. 2020 Jul 31;11:1825. doi: 10.3389/fpsyg.2020.01825. eCollection 2020. PMID 32849076
- [Background] Tsepilov YA, Freidin MB, Shadrina AS, Sharapov SZ, Elgaeva EE, Zundert JV, Karssen Lcapital ES, Cyrillic, Suri P, Williams FMK, Aulchenko YS. Analysis of genetically independent phenotypes identifies shared genetic factors associated with chronic musculoskeletal pain conditions. Commun Biol. 2020 Jun 25;3(1):329. doi: 10.1038/s42003-020-1051-9. PMID 32587327
- [Background] Crofford LJ. Chronic Pain: Where the Body Meets the Brain. Trans Am Clin Climatol Assoc. 2015;126:167-83. PMID 26330672
- [Background] Diatchenko L, Fillingim RB, Smith SB, Maixner W. The phenotypic and genetic signatures of common musculoskeletal pain conditions. Nat Rev Rheumatol. 2013 Jun;9(6):340-50. doi: 10.1038/nrrheum.2013.43. Epub 2013 Apr 2. PMID 23545734
- [Background] Kalkman JC, Visser K, Moen J, Bonsel JG, Grobbee ED, Moons MKG. Preoperative prediction of severe postoperative pain. Pain. 2003 Oct;105(3):415-423. doi: 10.1016/S0304-3959(03)00252-5. PMID 14527702
- [Background] Fillingim RB, King CD, Ribeiro-Dasilva MC, Rahim-Williams B, Riley JL 3rd. Sex, gender, and pain: a review of recent clinical and experimental findings. J Pain. 2009 May;10(5):447-85. doi: 10.1016/j.jpain.2008.12.001. PMID 19411059
- [Background] Wang L, Guyatt GH, Kennedy SA, Romerosa B, Kwon HY, Kaushal A, Chang Y, Craigie S, de Almeida CPB, Couban RJ, Parascandalo SR, Izhar Z, Reid S, Khan JS, McGillion M, Busse JW. Predictors of persistent pain after breast cancer surgery: a systematic review and meta-analysis of observational studies. CMAJ. 2016 Oct 4;188(14):E352-E361. doi: 10.1503/cmaj.151276. Epub 2016 Jul 11. PMID 27402075
- [Background] Theunissen M, Peters ML, Bruce J, Gramke HF, Marcus MA. Preoperative anxiety and catastrophizing: a systematic review and meta-analysis of the association with chronic postsurgical pain. Clin J Pain. 2012 Nov-Dec;28(9):819-41. doi: 10.1097/AJP.0b013e31824549d6. PMID 22760489
- [Background] Hinrichs-Rocker A, Schulz K, Jarvinen I, Lefering R, Simanski C, Neugebauer EA. Psychosocial predictors and correlates for chronic post-surgical pain (CPSP) - a systematic review. Eur J Pain. 2009 Aug;13(7):719-30. doi: 10.1016/j.ejpain.2008.07.015. Epub 2008 Oct 25. PMID 18952472
- [Background] Meretoja TJ, Andersen KG, Bruce J, Haasio L, Sipila R, Scott NW, Ripatti S, Kehlet H, Kalso E. Clinical Prediction Model and Tool for Assessing Risk of Persistent Pain After Breast Cancer Surgery. J Clin Oncol. 2017 May 20;35(15):1660-1667. doi: 10.1200/JCO.2016.70.3413. Epub 2017 Mar 13. PMID 28524782
- [Background] Fink R. Pain assessment: the cornerstone to optimal pain management. Proc (Bayl Univ Med Cent). 2000 Jul;13(3):236-9. doi: 10.1080/08998280.2000.11927681. PMID 16389388
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Lempa M, Koch G, Neugebauer E, Kohler L, Troidl H. [How much pain is tolerable? Target expectations of surgical patients for pain therapy]. Chirurg. 2000 Oct;71(10):1263-9. doi: 10.1007/s001040051213. German. PMID 11077589
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981
- [Background] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT06417528/Prot_SAP_000.pdf